CLINICAL TRIAL: NCT00292045
Title: Phase 1 Study of Immunization With NY-ESO-1 Protein Combined With CpG 7909 in Patients With High-risk Stage D1 or Advanced Prostate Cancer
Brief Title: Immunization With NY-ESO-1 Protein Combined With CpG 7909 in Patients With Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ludwig Institute for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUD2003-024; 2004DR1380 (SwissMedic); KEK-StV-Nr. 01/04 (local EC)
Record Dates: First submitted 2006-02-13; First posted 2006-02-15 (Estimated); Results first posted 2021-01-27 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Prostate Cancer
Keywords: NY-ESO-1 protein, immunization, advanced prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NY-ESO-1 protein + CpG 7909 (Experimental): Patients received immunization with intradermal injections of the NY-ESO-1 protein combined with CpG 7909.
  Interventions: Biological: NY-ESO-1 protein/CpG 7909

INTERVENTIONS:
Biological: NY-ESO-1 protein/CpG 7909 — Patients received vaccinations consisting of the NY-ESO-1 protein (100 µg) combined with CpG 7909 (2.5 mg) as an adjuvant administered intradermally every 3 weeks for 4 doses (i.e., 12-week cycle).

SUMMARY:
This was a Phase 1, open-label, fixed-dose study of immunization with the NY-ESO-1 protein combined with CpG 7909 as an adjuvant in patients with histopathologically confirmed, high-risk Stage D1 or advanced prostate cancer. The primary study objective was to assess the safety of NY-ESO-1 protein/CpG 7909 immunization, and the secondary objective was to evaluate the immunity induced by immunization.

DETAILED DESCRIPTION:
Eligible patients received vaccinations consisting of the NY-ESO-1 protein (100 µg) combined with CpG 7909 (2.5 mg) administered intradermally every 3 weeks for 4 doses. Patients who demonstrated stable disease, minor response, partial response, or complete response at Week 13 may have continued to receive vaccinations until disease progression. In patients with mixed response, single progressive lesions may have been resected and vaccination may have been continued.

Safety was monitored continuously. Blood samples were obtained for clinical hematology, biochemistry and immune response assessments, including antinuclear antibody (ANA) and anti-dsDNA, NY-ESO-1 and/or LAGE-1 specific antibodies, and NY-ESO-1 specific cluster of differentiation (CD)4+ and CD8+ T cells.

A tumor sample, resected prior to immunization, was tested to determine NY-ESO-1 and/or LAGE-1 expression. Delayed-type hypersensitivity (DTH) testing was performed at baseline and on study.

Disease status was assessed at baseline and on study in patients with measurable disease.

ELIGIBILITY:
Inclusion Criteria

Patients were eligible for enrollment if they fulfilled the following criteria:

1. High-risk Stage D1 or metastatic prostate cancer (D2), confirmed by review of histology.
2. Fully recovered from surgery.
3. Showed stable or progressive disease as assessed by X-ray, ultrasound, and/or computed tomography (CT) scans under hormonal and/or chemotherapeutic treatment, which had been administered for ≥ 3 months.
4. Any pretreatment with chemo- or radiotherapy must have been discontinued for ≥ 4 weeks prior to the first dose of study agent. Hormone therapy was allowed before and throughout the study.
5. Expected survival of ≥ 3 months.
6. Karnofsky performance status of ≥ 70%.
7. Within the last 2 weeks prior to study day 1, vital laboratory parameters should have been within the normal range, except for the following laboratory parameters, which should have been within the ranges specified:

   * Leukocytes > 3,000/µl.
   * Lymphocytes > 700/µl.
   * Platelets > 100,000/µl.
   * Serum creatinine < 2.5 mg/dL.
   * Alanine aminotransferase, aspartate aminotransferase, and total bilirubin < 2.5 x upper limit of normal.
8. Age ≥ 18 years.
9. Able to give valid written informed consent.

Exclusion Criteria

Patients were excluded from the study if they fulfilled any of the following criteria:

1. Clinically significant heart disease (i.e., New York Heart Association Class 3 congestive heart failure; myocardial infarction within the past 6 months; unstable angina; coronary angioplasty within the past 6 months; uncontrolled atrial or ventricular cardiac arrhythmias).
2. Other serious illnesses, e.g., active infections requiring antibiotics, bleeding disorders.
3. Concomitant systemic treatment with corticosteroids. Topical or inhalational steroids were permitted.
4. Metastatic disease to the central nervous system.
5. Mental impairment, in the opinion of the Investigator, that may have compromised the ability to give informed consent and comply with the requirements of the study.
6. Lack of availability for immunological and clinical follow-up assessments.
7. Participation in chemotherapy, radiation therapy, or any other clinical trial involving another investigational agent within 4 weeks prior to first dosing.
8. Being a recipient of an organ or bone marrow allograft. Having an autoimmune disease other than vitiligo, such as, but not limited to, inflammatory bowel disease or multiple sclerosis.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2004-10-27 (Actual); Primary Completion 2006-01-09 (Actual); Study Completion 2006-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Knuth, MD, Principal Investigator — Clinic of Oncology, University Hospital Zürich, Switzerland; Elke Jäger, MD, PhD, Principal Investigator — II. Medizinische Klinik, Hämatologie/Onkologie, Krankenhaus Nordwest, Frankfurt
Locations (2):
- Krankenhaus Nordwest, Frankfurt, Germany
- Universitätsspital Zürich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Therasse P, Arbuck SG, Eisenhauer EA, Wanders J, Kaplan RS, Rubinstein L, Verweij J, Van Glabbeke M, van Oosterom AT, Christian MC, Gwyther SG. New guidelines to evaluate the response to treatment in solid tumors. European Organization for Research and Treatment of Cancer, National Cancer Institute of the United States, National Cancer Institute of Canada. J Natl Cancer Inst. 2000 Feb 2;92(3):205-16. doi: 10.1093/jnci/92.3.205. PMID 10655437
- [Result] Karbach J, Neumann A, Atmaca A, Wahle C, Brand K, von Boehmer L, Knuth A, Bender A, Ritter G, Old LJ, Jager E. Efficient in vivo priming by vaccination with recombinant NY-ESO-1 protein and CpG in antigen naive prostate cancer patients. Clin Cancer Res. 2011 Feb 15;17(4):861-70. doi: 10.1158/1078-0432.CCR-10-1811. Epub 2010 Dec 16. PMID 21163871

RESULTS

PARTICIPANT FLOW:
Groups:
- NY-ESO-1 Protein + CpG 7909: Patients received vaccinations consisting of the NY-ESO-1 protein (100 µg) combined with CpG 7909 (2.5 mg) as an adjuvant administered intradermally every 3 weeks for 4 doses (i.e., 12-week cycle). Patients who demonstrated stable disease, minor response, partial response, or complete response at Week 13 may have continued to receive vaccinations until disease progression.
Period: Core Study (Through Week 13)
Arm/Group | NY-ESO-1 Protein + CpG 7909
Started | 15
Completed (Completion of Cycle 1 (4 vaccinations given once every 3 weeks, for a total cycle length of 12 weeks) plus 3 weeks of follow-up) | 13
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Period: Extended Treatment Beyond Week 13
Arm/Group | NY-ESO-1 Protein + CpG 7909
Started | 10
Completed (Completion of extended treatment was not defined; patients received between 1 and 4 vaccinations during extended treatment (in addition to the 4 vaccinations in the Core Study)) | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The population comprises all enrolled patients.
Arm/Group | NY-ESO-1 Protein + CpG 7909
Number analyzed (Participants) | 15
Age, Continuous [Median (Full Range); unit: years] | 67 [46 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Switzerland | 3
  Germany | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Treatment-emergent Adverse Events (TEAEs)
Description: Toxicity was graded in accordance with the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 3.0, as follows: Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe), Grade 4 (life-threatening), and Grade 5 (fatal). Adverse events (AEs) were reported based on clinical laboratory tests, vital sign and weight measurements, physical examinations, performance status evaluations, and any other medically indicated assessments, including patient interviews, from the first dose of study treatment through the final follow-up visit. AEs were considered to be treatment emergent (TEAE) if they occurred or worsened in severity after the first dose of study treatment.
Time Frame: Up to 56 weeks
Population: The population comprises all patients who received any dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | NY-ESO-1 Protein + CpG 7909
Number analyzed (Participants) | 15
Participants
  Any TEAE | 15
  Maximum TEAE severity Grade 1 | 2
  Maximum TEAE severity Grade 2 | 10
  Maximum TEAE severity Grade 3 | 2
  Maximum TEAE severity Grade 4 | 1
  Serious TEAE | 4
  TEAE leading to discontinuation | 1

2. Secondary Outcome: Number of Patients With Cellular Antibody Response to NY-ESO-1
Description: Assays to assess cluster of differentiation (CD)4+ and CD8+ antigen-specific responses were performed at baseline (within 14 days prior to the first vaccination) and during the vaccination period (Weeks 4, 10, 16, 22, and 28) by enzyme-linked immune absorbent spot (ELISPOT) assay. A positive response was considered if the number of spots in the peptide-exposed well was 2-fold or more higher than the number of spots in the unstimulated well, and if there was a minimum of 10 (after subtraction of background spots) peptide-specific spots/25.000 T cells or less if T-cell clones were used.
Time Frame: Up to 28 weeks
Population: The population comprises all patients who received at least 4 vaccinations with study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | NY-ESO-1 Protein + CpG 7909
Number analyzed (Participants) | 13
Participants
  CD4+ T cell response | 9
  CD8+ T cell response | 6

3. Secondary Outcome: Number of Patients With Humoral Antibody Response to NY-ESO-1
Description: Assays to assess NY-ESO-1 specific antibodies were performed at baseline (within 14 days prior to the first vaccination) and during the vaccination period (Weeks 4, 7, 10, 13, 16, 19, 22, 25, and 28). Sera were assessed over a range of dilutions from 1:100 to 1:400,000. Vaccine-induced antibodies were mapped with a panel of overlapping 20 mer peptides (25 μg/mL) spanning the whole protein sequence by enzyme-linked immunosorbent assay (ELISA). Immunoglobulin (Ig) subclasses G1 and G3 were determined by Western blot analysis using secondary antibody mouse anti-human IgG1/IgG3 at a dilution of 1:1000.
Time Frame: Up to 28 weeks
Population: The population comprises all patients who received at least 4 vaccinations with study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | NY-ESO-1 Protein + CpG 7909
Number analyzed (Participants) | 13
Participants | 13

4. Secondary Outcome: Number of Patients With Best Tumor Response as Measured by the Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Appropriate imaging scans were performed at baseline (within 14 days prior to the first vaccination) and during the vaccination period (Weeks 13 and 28). Response was assessed using RECIST version 1.0 (Therasse et al, J Natl Cancer Inst 2000; 92:205-16). Per RECIST, target lesions are categorized as follows: complete response (CR): disappearance of all target lesions (no evaluable disease); partial response (PR): ≥ 30% decrease in the sum of the longest diameter of target lesions; progressive disease (PD): ≥ 20% increase in the sum of the longest diameter of target lesions; stable disease (SD): small changes that do not meet above criteria.
Time Frame: Up to 32 weeks
Population: The population comprises all patients who received at least 4 vaccinations with study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | NY-ESO-1 Protein + CpG 7909
Number analyzed (Participants) | 13
Participants
  Stable disease | 8
  Progressive disease | 3
  No evidence of disease at baseline and on study | 2

ADVERSE EVENTS:
Time Frame: All adverse events (AEs), regardless of causality to study drug, were documented from the first dose of study treatment through the final follow-up visit, for an AE collection period of up to 56 weeks for each patient.
Description: AE documentation included onset/resolution dates, severity using the NCI CTCAE (version 3.0), seriousness, relationship to study drug, study drug action taken, treatment, and outcome. In summaries, preferred terms were counted only once per patient at the maximum reported grade.
Arm/Group | NY-ESO-1 Protein + CpG 7909
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 4/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NY-ESO-1 Protein + CpG 7909 (N=15)
Paraplegia (Nervous system disorders) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Hypotension (Vascular disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Oedema peripheral (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NY-ESO-1 Protein + CpG 7909 (N=15)
Bradycardia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Accommodation disorder (Eye disorders) | 1
Eye irritation (Eye disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Injection site erythema (General disorders) | 13
Pyrexia (General disorders) | 12
Influenza like illness (General disorders) | 4
Chills (General disorders) | 3
Injection site pain (General disorders) | 2
Injection site vesicles (General disorders) | 2
Oedema peripheral (General disorders) | 1
Asthenia (General disorders) | 1
Feeling cold (General disorders) | 1
Injection site necrosis (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Urinary tract infection (Infections and infestations) | 3
Tooth infection (Infections and infestations) | 1
Weight decreased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
C-reactive protein increased (Investigations) | 1
Karnofsky scale worsened (Investigations) | 1
Weight increased (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 4
Sciatica (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Sleep disorder (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 2
Nocturia (Renal and urinary disorders) | 2
Pollakiuria (Renal and urinary disorders) | 2
Bladder pain (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 1
Skin maceration (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 2
Deep vein thrombosis (Vascular disorders) | 1
Hot flush (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less